CLINICAL TRIAL: NCT03968835
Title: A Comparison of the Outcomes of Distal Fingertip Amputations Treated With Either Artificial (Xeroform) or Biological Dressings
Status: Withdrawn | Type: Observational
Why Stopped: lack of enrollment
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Other Study IDs: 18-00132
Record Dates: First submitted 2019-05-08; First posted 2019-05-30 (Actual); Last update posted 2020-05-29 (Actual); Status verified 2020-05

CONDITIONS: Finger Injuries; Amputation, Traumatic
MeSH Terms: conditions — Finger Injuries; Amputation, Traumatic | interventions — Bacitracin; Skin Transplantation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Biological Dressings: Bacitracin will be applied and covered with xeroform and gauze
  Interventions: Other: Bacitracin
- Artificial Dressings: the amputated composite skin and soft tissue unit will be thinned out to become a full thickness skin graft
  Interventions: Other: Skin Graft

INTERVENTIONS:
Other: Bacitracin — For the first 30 people, bacitracin will be applied and covered with xeroform and gauze.
  Groups: Biological Dressings
Other: Skin Graft — For the next 30 patients, the amputated composite skin and soft tissue unit will be thinned out to become a full thickness skin graft.
  Groups: Artificial Dressings

SUMMARY:
This is a prospective study looking to evaluate whether the treatment outcomes for patients who sustain a distal fingertip amputation are improved or no different when using biological dressings versus artificial dressings.

ELIGIBILITY:
Inclusion Criteria:

* All individuals presenting at Bellevue Hospital for evaluation and treatment of a finger amputation distal to the germinal matrix that present along with the amputated distal fingertip unit.

Exclusion Criteria:

* replantation candidate, incomplete distal finger-tip amputation

Max Age: 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: 60 patients will be followed for the study. The first 30 patients will be treated with biological dressings and subsequent 30 patients will be treated with artificial dressings.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2018-12-24 (Actual); Primary Completion 2021-05 (Estimated); Study Completion 2021-05 (Estimated)

PRIMARY OUTCOMES:
Time to complete healing up to 3 Months | 3 months
Percentage of graft viability (for biological dressing only) | 1 week
Percentage of graft viability (for biological dressing only) | 3 weeks
Percentage of graft viability (for biological dressing only) | 6 weeks
Percentage of graft viability (for biological dressing only) | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Jacques Hacquebord, Principal Investigator — New York Langone Medical Center
Locations (1):
- New York University School of Medicine, New York, New York, United States